CLINICAL TRIAL: NCT05019300
Title: Long-term Neurocognitive and Psychiatric Consequences of COVID-19 in Patients Discharged From Critical Care Units. A Cohort Study of the Advance Interdisciplinary Rehabilitation Register (AIRR) Covid-19 Working Group.
Brief Title: Long-term Neurocognitive and Psychiatric Consequences in Severe COVID-19 Survivors.
Acronym: NPQCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Constanza Caneo, Clinical Assistant Professor, C-L Psychiatrist, PI NPQCOVID, Advance Interdisciplinary Rehabilitation Register, (AIRR) Covid-19 Working group, Pontificia Universidad Catolica de Chile
Other Study IDs: 0000001; 1U19AI135972 (NIH)
Record Dates: First submitted 2021-08-20; First posted 2021-08-24 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Neurocognitive Dysfunction
Keywords: COVID-19; Intensive Care Units; Functionality; Fatigue; Anxiety; Insomnia; Long-term cognitive impairment; language disorders; Verbal fluency; Depression; Post traumatic stress; exercise endurance
MeSH Terms: conditions — COVID-19; Cognition Disorders; Fatigue; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Language Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients discharged from critical care units: Adults over 18 years of age who have been hospitalized after COVID-19 diagnosis in the critical care units of Red Salud UC Christus who have been cognitively evaluated with Montreal Cognitive Assessment (MoCA) days prior to their discharge. All patients with a previous history of confirmed neurocognitive or psychotic disorders, prior to hospital admission, were excluded.
  Interventions: Biological: Exposure: COVID-19 severity

INTERVENTIONS:
Biological: Exposure: COVID-19 severity — COVID-19 severity between 4 to 7 points according the seven-category scale of clinical status reported by Huang et al. (2021) and severe to critical symptomatic levels on spectrum of disease reported by Wu and McGoogan (2020).

SUMMARY:
Long-term neurocognitive and psychiatric consequences of COVID-19 remain mostly unknown to date. It has been reported that coronaviruses cause direct central nervous system infection (Needham et al. 2020). Besides that, new or worsening cognitive impairment commonly occurs and persists in survivors of intensive care unit (ICU) stay (Hosey & Needham. 2020). The purpose of our study is to search and describe the cognitive and psychiatric long-term consequences of COVID-19 on patients who have been discharged from critical care units. This is an ambidirectional cohort study, that attempts to follow adults discharged from critical Care Units Adults due to COVID-19 up to 12 months after discharge, to evaluate the presence of cognitive impairment, linguistic and phonation function, depression, fatigue, functional gastroenterological symptoms, anxiety, or post traumatic disorder, and performance in activities of daily living and physical response to exercise as well.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age who have been hospitalized at critical care units, who were admitted for a diagnosis of COVID-19 and who present a score on the MOCA® cognitive test of less than 26 points at the time of hospital discharge .

Exclusion Criteria:

* History of underlying cognitive disorder. History of underlying primary psychotic disorder. MOCA® cognitive test score greater than or equal to 26 points at the time of hospital discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients over 18 years of age discharged from critical care units at Red de Salud UC Christus who presented MoCA® cognitive test result less than 26 points at the time of discharge.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment screening | 12 months
  Montreal Cognitive Assessment (MoCA®). Evaluation of cognitive domains (visuospatial, executive function; attention and memory; orientation; language).
  Min score: 0 Max score: 30 Cut-off for chilean population: < 21 for mild cognitive impairment. < 20 for dementia
  Setting: Home and online

SECONDARY OUTCOMES:
Cognitive performance | 12 months
  Cambridge Neuropsychological Test Automated Battery (CANTAB®)
  Included tests:
  Reaction time test, (RTI) Paired associate learning (PAL) Spatial Working Memory (SWM) Spatial Span (SSP) Rapid Visual Information Processing (RVP) Cambridge Gambling Task (CGT) Intra/Extra Dimensional Set Shift (IED) Stockings of Cambridge (SOC)
  Scores: z-scores normalized by sex and educational level
  Setting: Home
Neurological Soft Signs | 12 months
  Test: Heidelberg Neurological Soft Signs Scale
  16 items on five factors ("motor coordination": Ozeretzki's test, diadochokinesis, pronation/supination, finger-to-thumb opposition, speech and articulation; "sensory integration": gait, tandem walking, two-point discrimination; "complex motor tasks": finger-to-nose test, fist-edge-palm test; "right/left and spatial orientation": right/left orientation, graphesthesia, face-hand test, stereognosis; "hard signs": arm holding test, mirror movements). All items except for gait, tandem gait, Ozeretzki's test, speech and articulation and right/left orientation are assessed separately for both, right and left sites respectively. Ratings are given on a 0-3 point scale (no/slight/moderate/marked abnormality).
  Higher scores mean worse outcomes. Min score: 0 Max score: 48 No cut-off point established in the literature.
  Setting: Home
Anxiety | 12 months
  Test: Generalized Anxiety Disorder-7 score
  The seven items assess (1) feeling nervous, anxious, or on edge; (2) being able to stop or control worrying; (3) worrying too much about different things; (4) trouble relaxing; (5) being restless; (6) becoming easily annoyed or irritable; and (7) feeling afraid as if something awful might happen.
  Increasing scores on the scale are strongly associated with multiple domains of functional impairment and increasing anxiety.
  The cut-off point suggested is of ≥10 Min score: 0 Max score: 21
  Setting: online
Depressive syndrome | 12 months
  Test: Patient Health Questionary-2 (PHQ-2) score for screening of depressive syndrome
  The cut-off point suggested is of ≥3 Min score: 0 Max score: 6
  Setting: online
Post Traumatic Stress Disorder | 12 months
  Test: Post Traumatic Checklist for Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) score
  20-item self-report measure that assesses the 20 DSM-5 symptoms of Post Traumatic Stress Disorder.
  The cut-off point suggested is of ≥33 Min score: 0 Max score: 80
  Setting: online
Physical disability | 12 months
  Test: Barthel Index score
  Measures physical disability behaviour relating to activities of daily living.
  Scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.
  Setting: online
Exercise endurance | 12 months
  Performance on 6 minutes- walk test
  Evaluation of aerobic capacity and exercise endurance.
  Setting: Home
Fatigue | 12 months
  Measured by the Modified fatigue impact scale (MFIS). The MFIS is a modified version of the 40-item Fatigue Impact Scale (FIS), which was originally developed to assess the effects of fatigue on quality of life in patients with chronic diseases. The FIS has patients rate the extent to which fatigue has affected their life in the past 4 weeks on a questionnaire consisting of 10 "physical" items, 10 "cognitive" items, and 20 "social" items, with 0 indicating "no problem" and 4 indicating "extreme problem."
  The cut-off point suggested is of ≥38 Min score: 0 Max score: 160
  Setting: online
Global functionality | 12 months
  Post-Covid-19 functional scale 5 levels of severity, where o is non impairment and 5 is the highest level of impairment.
  Setting: online
Quality of life related to health | 12 months
  Test: The 5-level EuroQol 5D health questionnaire. (EQ-5D-5L) Self rated.
  Min score: 0 Max score: 100 highest score means worst quality of life.
  Setting: online
Muscle strength | 12 months
  Dynamometry Setting: Home
Pain severity | 12 months
  Scale: Stanford pain scale
  Min: 0 represents no pain Max: 10 represents unimaginable or unspeakable pain Setting: online
Spontaneous Speech | 12 months
  Spontaneous Speech is a useful research tool to assess the scope of language disorders in people with neurological deficits. Short samples be analyzed during a brief interview and based of 10 linguistics parameters, it will characterized level and the type of language deficit. The 10 linguistic parameters are based on the ALEA method
  Setting: Home and online
Verbal fluency | 12 months
  Verbal fluency (phonological and sematic) will be assed by requesting the participants to elicit word under 1 minute for letter F, A and S and for the category animals.
  Setting: Home and online
complex post-traumatic stress disorder | 12 months
  Test: International Trauma Questionnaire self-report measure for post-traumatic stress disorder (PTSD) and complex post-traumatic stress disorder (CPTSD), corresponding to the diagnostic criteria in the International Classification of Diseases, 11th Revision (ICD-11).
  Setting: online
irritable bowel syndrome | 12 months
  Rome IV criteria Setting: online
Insomnia | 12 months
  Scale: Pittsburgh insomnia rating scale
  Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
  Setting: online
Dysautonomia | 12 months
  Scales: Scales for outcomes in Parkinson's dysfunction-autonomic (SCOPA-AUT), Orthostatic hypotension symptom assessment (OHSA) and Orthostatic hypotension activity scale (OHACT).
  Setting: online
Dyspnea | 12 months
  Test: Chronic obstructive pulmonary disease (COPD) assessment test (CAT).
  Min: 0 Max: 40 CAT ≥10 corresponds to either GOLD Group B or D. Group B patients' preferred treatment is to start either on LABA, or LAMA and if persistent symptoms then combination LAMA/LABA therapy-these are the minimum for patients with CAT Score ≥10.
  CAT <10 corresponds to GOLD Group A or C. Group A patients' preferred treatment is to start bronchodilator (LABA or LAMA) and evaluate the effect.
  Setting: online

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Medina, PhD, Study Director — Pontificia Universidad Catolica de Chile; Arnoldo Riquelme, PhD, Study Director — Pontificia Universidad Catolica de Chile; Constanza Caneo, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Carolina Mendez, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Investigaciones Médicas, Centro de Investigación Clínica UC, Hospital Clínico UC, San Carlos de Apoquindo, Departamento de Ciencias de la Salud, Escuela de Medicina, Red UC-Christus, Campus Clínico San JoaPontificia Universidad Catolica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
We are available to be contacted by researchers aiming to conduct secondary analyses based on our study, after providing a study protocol based on international guidelines, in order to ensure adequate use of our data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2024
Access Criteria: contact to responsable researcher C Caneo

REFERENCES:
- [Background] Hosey MM, Needham DM. Survivorship after COVID-19 ICU stay. Nat Rev Dis Primers. 2020 Jul 15;6(1):60. doi: 10.1038/s41572-020-0201-1. PMID 32669623
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Kotfis K, Williams Roberson S, Wilson JE, Dabrowski W, Pun BT, Ely EW. COVID-19: ICU delirium management during SARS-CoV-2 pandemic. Crit Care. 2020 Apr 28;24(1):176. doi: 10.1186/s13054-020-02882-x. PMID 32345343
- [Background] Oxley TJ, Mocco J, Majidi S, Kellner CP, Shoirah H, Singh IP, De Leacy RA, Shigematsu T, Ladner TR, Yaeger KA, Skliut M, Weinberger J, Dangayach NS, Bederson JB, Tuhrim S, Fifi JT. Large-Vessel Stroke as a Presenting Feature of Covid-19 in the Young. N Engl J Med. 2020 May 14;382(20):e60. doi: 10.1056/NEJMc2009787. Epub 2020 Apr 28. No abstract available. PMID 32343504
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Needham EJ, Chou SH, Coles AJ, Menon DK. Neurological Implications of COVID-19 Infections. Neurocrit Care. 2020 Jun;32(3):667-671. doi: 10.1007/s12028-020-00978-4. PMID 32346843
- [Background] Alberti P, Beretta S, Piatti M, Karantzoulis A, Piatti ML, Santoro P, Vigano M, Giovannelli G, Pirro F, Montisano DA, Appollonio I, Ferrarese C. Guillain-Barre syndrome related to COVID-19 infection. Neurol Neuroimmunol Neuroinflamm. 2020 Apr 29;7(4):e741. doi: 10.1212/NXI.0000000000000741. Print 2020 Jul. No abstract available. PMID 32350026
- [Background] Toscano G, Palmerini F, Ravaglia S, Ruiz L, Invernizzi P, Cuzzoni MG, Franciotta D, Baldanti F, Daturi R, Postorino P, Cavallini A, Micieli G. Guillain-Barre Syndrome Associated with SARS-CoV-2. N Engl J Med. 2020 Jun 25;382(26):2574-2576. doi: 10.1056/NEJMc2009191. Epub 2020 Apr 17. No abstract available. PMID 32302082
- [Background] Solomon T. Neurological infection with SARS-CoV-2 - the story so far. Nat Rev Neurol. 2021 Feb;17(2):65-66. doi: 10.1038/s41582-020-00453-w. PMID 33414554
- [Background] Valderrama EV, Humbert K, Lord A, Frontera J, Yaghi S. Severe Acute Respiratory Syndrome Coronavirus 2 Infection and Ischemic Stroke. Stroke. 2020 Jul;51(7):e124-e127. doi: 10.1161/STROKEAHA.120.030153. Epub 2020 May 12. No abstract available. PMID 32396456
- [Background] Beyrouti R, Adams ME, Benjamin L, Cohen H, Farmer SF, Goh YY, Humphries F, Jager HR, Losseff NA, Perry RJ, Shah S, Simister RJ, Turner D, Chandratheva A, Werring DJ. Characteristics of ischaemic stroke associated with COVID-19. J Neurol Neurosurg Psychiatry. 2020 Aug;91(8):889-891. doi: 10.1136/jnnp-2020-323586. Epub 2020 Apr 30. No abstract available. PMID 32354768